CLINICAL TRIAL: NCT05765097
Title: Clinical Application of an Open-source Artificial Pancreas System in Adult Inpatients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xuefeng Yu, Professor, Chief Physician，Director of Department of Endocrinology, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZRKY-2022-01
Record Dates: First submitted 2023-02-08; First posted 2023-03-13 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study was conducted in two phases: one subject only participated in one of the phases.
  In phase 1, the semi-closed-loop open source AP system was used to treat the subjects, and the nurse manually entered the initial basal and the bolus instruction for three meals into the system according to the doctor's advice. When the Phase 1 trial is completed, all subjects have no serious adverse events and have been evaluated and confirmed by participants, the phase 2 trial can proceed. In phase 2, the full closed-loop open source AP system was used to treat the subjects. The nurses manually entered initial basal into the system according to the doctor's advice to start treatment, and the open source AP system automatically gave infusion instructions for boluses.Each phase will enroll up to 10 subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artificial pancreas group (Experimental): Using artificial pancreas system (composed of a CGM, a pump and AndroidAPS software) to treat adult patients with diabetes
  Interventions: Device: Artificial pancreas treatment

INTERVENTIONS:
Device: Artificial pancreas treatment — five to seven days treatment by artificial pancreas system

SUMMARY:
Open-source artificial pancreas system has been applied in clinical settings abroad for several years, and its safety and effectiveness has been reported by many literature. However, there is no reporting of its clinical application in China. Taking the inpatients with diabetes in the Department of Endocrinology as the starting point of research, participants would like to explore the safety and efficacy of open source artificial pancreas system in domestic clinical application, further to promote the development and landing of artificial pancreas technology in China, and finally to provide better treatment options for the majority of diabetes patients in China.

DETAILED DESCRIPTION:
Artificial Pancreas (AP), as the treatment of type 1 diabetes, has attracted more and more attention in recent years. The artificial pancreas system is an Automatic Insulin Delivery/AID device that consists of three main elements: The Continuous Glucose Monitoring , insulin pump and central algorithm control system ,it can automatically calculate the immediate insulin infusion dose according to the immediate blood glucose, giving continuous subcutaneous infusion, and maximizing the simulation of the physiological secretion pattern of human insulin, so as to achieve closed-loop blood glucose management. Compared with traditional insulin pump therapy , artificial pancreas system has advantages such as higher intelligence, more stable blood glucose control, and less burden of blood glucose management. While greatly improving patients' quality of life, its safety has also been verified in a number of foreign clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 18~75 years old (including 18 years old and 75 years old), gender is not limited;
2. Patients with type 1 diabetes mellitus (T1DM);
3. Patients with type 2 diabetes mellitus (T2DM) who require insulin therapy;
4. Those who sign the informed consent form and voluntarily participate in this clinical trial;
5. Be able to understand the trial and cooperate with the test procedure, and be able to follow up the observer as required.

Exclusion Criteria:

1. Patients who are not suitable for insulin pump therapy;
2. Acute complications of diabetes, such as diabetic ketoacidosis, diabetic hyperosmolar non-ketotic coma;
3. Hyperglycemia with severe circulatory disorders and patients with shock;
4. Cardiac function grade III or above; ALT or AST exceeds the upper limit of normal value by more than 3 times; Serum creatinine more than 442μmol/L; Hemoglobin less than 90g/L; White blood cell count < 4.0×109/L or platelet count <90×109/L;
5. Those who are allergic to adhesive tape;
6. Patients with skin diseases such as rash and prurigo, or abnormal coagulation function;
7. Women who are pregnant or lactating, or those who have a family plan during clinical trials;
8. Those who suffer from mental illness, have no self-control, and cannot express themselves clearly;
9. Those who have participated in clinical studies of other drugs, biologics or medical devices before screening but have not reached the time limit of the primary research endpoint;
10. Other circumstances that participants deems inappropriate to participate in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
TIR | 5-7days
  Time in range

SECONDARY OUTCOMES:
mean BG | 5-7 days
  mean blood glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China